CLINICAL TRIAL: NCT03723174
Title: Impact of an Educational Program on Oral Health Related Quality of Life in a Group of 11 to 14 Years Old Egyptian Children: Before and After Study.
Brief Title: Impact of an Educational Program on Gingival Status and Oral Health Related Quality of Life
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fayrouz Saber, Assistant lecturer, Cairo University
Other Study IDs: fay
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Gingival Disease; Oral Disease
MeSH Terms: conditions — Gingival Diseases; Mouth Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm: baseline data will be calculated before the oral health educational program using gingival index and after 3 months from the intervention
  Interventions: Behavioral: Oral Health Educational Program

INTERVENTIONS:
Behavioral: Oral Health Educational Program — proper introduction to brushing techniques, dietary recommendations and importance of visiting the dentist

SUMMARY:
This research targets the evaluation of the impact of oral health educational programs on the gingival status and oral health related quality of life in early adolescence of the Egyptian population. Each participant will benefit from the education of the proper oral hygiene practices under the supervision and follow up of the investigator in addition to the potential improvement of his/ her oral health related quality of life.

DETAILED DESCRIPTION:
The objective of this study is to improve the gingival status and oral health related quality of life in the Egyptian population's early adolescence. The intervention is an Oral health educational program based on the following:

* Tooth brushing: the modified bass technique is the method of choice the skill will be taught using a video followed by a model demonstration then a supervised brushing session done by the participants.
* Dietary recommendations and importance of visiting the dentist will be introduced in the form of power point presentation that will be set according to the American Academy of Pediatric Dentistry (AAPD).
* Participant will be asked to come for 4 visits one for base line data collection and administration of the intervention and another 3 follow up visits once per month.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged from 11-14 years old
2. No reported systemic disease
3. No administration of antibiotics in the last month
4. No fixed or removable appliance
5. Absence of acute phase of any oral disease

Exclusion Criteria:

1. Patient refuses to participate in the study
2. patient fails to attend follow up sessions

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged from 11 to 14 years old seeking dental care at the educational hospital, Department of Pediatric Dentistry and Dental Public Health, School of Dentistry New Giza University.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Short form Child perception questionnaire 11-14 | 3 months
  assessment of Oral symptoms, functional limitations, emotional and social well being. each domain scores from 0-20 where 20 means the worst quality of life in each domain.

SECONDARY OUTCOMES:
Photographic evaluation and interpretation using Adobe Photoshop Creative Cloud 2021 | 3 months
  assessment of Swelling of gingiva red color characteristics using number of red pixels

CONTACTS AND LOCATIONS:
Overall Officials: Manal Al Sayed, PhD, Study Director — Professor
Locations (1):
- New Giza University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhardwaj VK, Sharma KR, Luthra RP, Jhingta P, Sharma D, Justa A. Impact of school-based oral health education program on oral health of 12 and 15 years old school children. J Educ Health Promot. 2013 Jul 31;2:33. doi: 10.4103/2277-9531.115820. eCollection 2013. PMID 24083283
- [Background] Smith RN, Lath DL, Rawlinson A, Karmo M, Brook AH. Gingival inflammation assessment by image analysis: measurement and validation. Int J Dent Hyg. 2008 May;6(2):137-42. doi: 10.1111/j.1601-5037.2008.00294.x. PMID 18412727
- [Result] Mostafa B, El-Refai I. Prevalence of Plaque-Induced Gingivitis in a Sample of the Adult Egyptian Population. Open Access Maced J Med Sci. 2018 Mar 10;6(3):554-558. doi: 10.3889/oamjms.2018.131. eCollection 2018 Mar 15. PMID 29610619